CLINICAL TRIAL: NCT01406028
Title: Does Emotional Support During the Luteal Phase Decrease the Stress of IVF?
Brief Title: Does Emotional Support Decrease In Vitro Fertilization Stress?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Rachel K. Ashby, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2009p-001214
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: In Vitro Fertilization; Psychological Stress
Keywords: IVF; Stress; Infertility
MeSH Terms: conditions — Stress, Psychological; Infertility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Standard of care includes discharge instructions from one of our IVF nurses regarding medications and timing of follow-up, at which point patients are told what day they need to return for their pregnancy test. Patients have access to phone numbers for their IVF nurses and physicians, as well as information about how to contact the social workers if additional support is needed. They also are provided the emergency phone numbers for after-hour calls to the fellow on call. However, during the time between the embryo transfer and the pregnancy test, the current standard of care is that contact between the patient and our team is patient-initiated.
- Intervention phone calls (Active Comparator): The intervention consisted of two phone calls from an IVF social worker during the time between embryo transfer and pregnancy test. The first phone call occurred between days 2-4 after transfer and the second phone call occurred between days 5 and 9 after embryo transfer. Standard language for introductions to phone calls and for voice mails was established prior to the start of the study.
  Interventions: Behavioral: Phone calls

INTERVENTIONS:
Behavioral: Phone calls — Phone calls to offer emotional support
  Arms: Intervention phone calls

SUMMARY:
In vitro fertilization for infertility has been associated with a significant amount of treatment related stress for patients. In addition,stress levels increase between embryo transfer and pregnancy test, during this waiting period. The investigators evaluated whether or not brief interventions by phone by trained social workers influenced stress levels. Our data showed that these interventions did not change levels, but confirmed that stress did increase during this time and that patients report wanting additional emotional support to improve stress during this period.

ELIGIBILITY:
Inclusion Criteria:

* All women (ages 18-45) undergoing their first fresh cycle of IVF using autologous oocytes where an embryo transfer occurred

Exclusion Criteria:

* > 2nd cycle of IVF IVF using donor eggs or a gestational carrier
* Transfers with Cryopreserved embryos
* Day 5 embryo transfers
* Self-reported history of depression or anxiety
* Already seeing a mental health professional
* Inability to speak or read English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale Scores | Day of embryo transfer (day 1) and 10 days later
  The perceived stress scale is a validated instrument to assess psychological stress

SECONDARY OUTCOMES:
Patient perceived benefit | 10 days after embryo transfer
  Exit questionnaires were administered 10 days after transfer to assess patient perceptions of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States